CLINICAL TRIAL: NCT06586008
Title: The Association Between Visual Echocardiographic Scoring System and Clinical Outcomes in Patient With Acute Decompensated Heart Failure
Acronym: VISCO-HF
Status: Recruiting | Type: Observational
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Sodiqur Rifqi, Principal Investigator; Former of Head of Department of Cardiovascular Medicine Faculty of Medicine Universitas Diponegoro, Universitas Diponegoro
Other Study IDs: Undip_Kardio 3
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Decompensated Heart Failure
Keywords: visual echocardiographic system; acute decompensated heart failure; mortality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the association between visual echocardiographic scoring system (visual mitral and tricuspid = VMT score) with clinical outcome among patients with acute decompensated heart failure. Researchers will collect information based on hospital registry as secondary data of in patient who had diagnosed as acute decompensated heart failure. The data consist of demographic data, clinical presentation, laboratory, and echocardiographic result were collected from hospital registry by reviewing medical record and echocardiographic machine database. Then, the data was analyzed by using IBM SPSS Statistics v26.

ELIGIBILITY:
Inclusion Criteria:

* Patient with history of heart failure with reduced ejection fraction (LVEF <40%)
* Age between 18 - 70 years old

Exclusion Criteria:

* Patient with pulmonary hypertension
* Patient with acute de novo heart failure (e.g. due to acute coronary syndrome)
* Significant valvular heart disease (more than moderate regurgitation or more than mild stenosis)
* Prior valve replacement/repair
* Patient with congenital heart disease
* Patient with pericardial disease
* Patient with poor echocardiographic images

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with acute decompensated heart failure who fulfill eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | During hospitalization, up to 1 weeks
  Mortality within hospitalization

SECONDARY OUTCOMES:
ICCU Length of Stay | During hospitalization, up to 1 weeks
Urine output | During hospitalization, up to 1 weeks
  24 hour urine output

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murayama M, Iwano H, Nishino H, Tsujinaga S, Nakabachi M, Yokoyama S, Aiba M, Okada K, Kaga S, Sarashina M, Chiba Y, Ishizaka S, Motoi K, Nishida M, Shibuya H, Kamiya K, Nagai T, Anzai T. Simple Two-Dimensional Echocardiographic Scoring System for the Estimation of Left Ventricular Filling Pressure. J Am Soc Echocardiogr. 2021 Jul;34(7):723-734. doi: 10.1016/j.echo.2021.02.013. Epub 2021 Mar 3. PMID 33675942
- [Background] Murayama M, Iwano H, Obokata M, Harada T, Omote K, Kagami K, Tsujinaga S, Chiba Y, Ishizaka S, Motoi K, Tamaki Y, Aoyagi H, Nakabachi M, Nishino H, Yokoyama S, Tanemura A, Okada K, Kaga S, Nishida M, Nagai T, Kurabayashi M, Anzai T. Visual echocardiographic scoring system of the left ventricular filling pressure and outcomes of heart failure with preserved ejection fraction. Eur Heart J Cardiovasc Imaging. 2022 Apr 18;23(5):616-626. doi: 10.1093/ehjci/jeab208. PMID 34694368